CLINICAL TRIAL: NCT05512975
Title: Evaluation of Protein Bioavailability, Satiety and Appetite Responses to Protein Fortified Porridge in Older Adults
Brief Title: FortiPhy: Protein Bioavailability, Satiety and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: The Norwegian Institute of Food, Fisheries and Aquaculture research (NOFIMA) (Unknown); National Research Institute for Agriculture, Food and environment (INRAE) (Unknown); Biotechnology and Biological Sciences Research Council (Other); European Joint Programming Initiative A Healthy Diet for a Healthy Life (JPI HDHL) (Unknown)
Responsible Party: Principal Investigator, Lisa Methven, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UREC 22/20
Record Dates: First submitted 2022-08-11; First posted 2022-08-23 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Protein-Energy Malnutrition
Keywords: Appetite; Older adults; Protein bioavailability; Satiety
MeSH Terms: conditions — Protein-Energy Malnutrition

STUDY DESIGN:
Intervention Model Description: Single group, cross-over design where each participant will consume one of 3 different porridge recipes on separate testing visits.
  The study will be conducted single blind as it not feasible to blind the researcher. Each participant will attend 3 study visits and all porridges will be provided in a blind manner.
Who Masked: Participant
Masking Description: Single blinded study. All participants will consume 2 fortified meals and 1 placebo/ control meal. All participants will be blinded to the intervention provided
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Porridge arm (Experimental): Control/ regular protein porridge recipe, not containing any additional protein fortification.
  Interventions: Dietary Supplement: Control Porridge arm
- Dairy Protein Porridge arm (Experimental): Porridge containing regular protein ingredients with dairy protein fortification (delical- a whey protein powder)
  Interventions: Dietary Supplement: Dairy protein porridge arm
- Plant Protein Porridge arm (Experimental): Porridge containing regular protein ingredients with plant protein fortification (extruded soy and soya milk)
  Interventions: Dietary Supplement: Plant protein porridge arm

INTERVENTIONS:
Dietary Supplement: Dairy protein porridge arm — Regular porridge ingredients with additional delical whey protein fortification
  Arms: Dairy Protein Porridge arm
Dietary Supplement: Plant protein porridge arm — Regular porridge ingredients with the addition of extruded soya protein fortification and soya milk instead of regular dairy milk
  Arms: Plant Protein Porridge arm
Dietary Supplement: Control Porridge arm — Regular porridge ingredients with no additional protein fortification
  Arms: Control Porridge arm

SUMMARY:
Older adults have very specific food and nutrient requirements and often struggle to meet these needs due to poor appetite, reduced functionality and dexterity. Protein (both quality and quantity) is an important macronutrient in maintaining muscle in older adults which can help prevent falls, delay disease onset and help individuals maintain independence. Fortifying regular/ everyday foods with additional protein is one strategy to help older adults meet these increased protein needs. However, it is well established that protein is the most satiating of the nutrients we eat, yet less is known about how this is impacted by age and protein type. This study aims to test 2 protein fortified porridge recipes in older adults (and a control recipe) with outcomes focused on protein bioavailability, appetite and satiety responses.

DETAILED DESCRIPTION:
Older adults have very specific food needs, not just in terms of the nutritional composition, but also because of reduced ability to prepare foods due to reduced functionality and dexterity. Foods may also become less appealing and less palatable with decreases in smell, taste and sight. Older adults often have a smaller appetite due to numerous factors including sensory decline, frailty, reduced activity and delayed gastric emptying. As such, fortified recipes of normal everyday foods can provide palatable familiar foods, that can be easy to prepare, whilst providing sufficient nutrients in a smaller portion size.

Within meals, the quality and quantity of dietary protein plays a significant role in maintaining muscle mass in older adults which can prevent falls and help older adults maintain their independence. Animal-based proteins (such as diary proteins) are complete protein sources that can lead to an improved muscle mass synthesis response compared to plant-based protein. However, it is also well established that protein is the most satiating of the nutrients we eat; yet less is known about how this is effected by age and by protein type. Hence, the addition of protein to a meal may result in an undesirable compensatory decrease in food intake in older adults, which may worsen undernutrition rather than preventing it. This issue is all the more worthwhile to investigate as ageing is known to alter hunger and satiety regulation mechanisms. Gastric emptying and gastrointestinal transit has been shown to delay in older adults. Slower gastric emptying can result in the stomach remaining distended a longer period of time and satiety being maintained. In addition, several studies have demonstrated the presence of higher levels of the hormones that control appetite in older compared to young individuals.

This study will be testing protein fortified porridge, a recipe that has been developed with older adults. It will assess how much of the protein in the meals is absorbed into the body and the impact it has on food intake, appetite, emptying from the stomach and hormones related to appetite. It will compare three recipes: a standard porridge recipe (control), a recipe fortified with milk protein (animal based protein), and a recipe fortified with soya (plant based protein).

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or over (no upper age limit), equal number of males and females
* BMI range: 18.5-30kg/m2
* Regularly consume 3 meals a day (with breakfast by 11am, lunch and dinner)
* Able to test the dishes provided
* Able to feed themselves
* Able to provide informed consent
* Understand English

Exclusion Criteria:

* Existing neurological or gastrointestinal condition
* Current chewing or swallowing difficulties (such as dysphagia)
* Existing cognitive or psychiatric disorder
* Taking medications that can significantly affect taste changes, appetite or gastric emptying
* On a special or therapeutic diet
* Have any food allergies or intolerances that will be worsened with meals provided in the study
* Have a history or drug or alcohol misuse
* Smoke more than 10 cigarettes a day
* Those who score ≤22 on the T-CogS exam

For participants providing blood samples:

* Anaemia (men: haemoglobin<130 g/L and women <115 g/L)
* Hypertension (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Protein Bioavailability: Do the dairy and soya protein fortified porridge recipes increase protein bioavailability in | 15-30 minute intervals for up to 4 hours following meal ingestion. This will be done for all 3 test meals provided to the participant
  Blood samples will be taken every 15-30 minutes following meal ingestion, and protein bioavailability will be determined in the samples using HPLC analysis.

SECONDARY OUTCOMES:
Appetite rating: Do the dairy and soya protein fortified recipes increase satiety and appetite responses in older adults compared to the non-fortified meals? | 30 minute intervals for up to 4 hours following meal ingestion. This will be done for all 3 test meals provided to the participant
  Appetite are assessed using a 100 mm Visual Analogue Scales (VAS, scale 0-100).

OTHER OUTCOMES:
Gastric emptying | 15-30 minute intervals for up to 4 hours following meal ingestion
  Gastric emptying is measured using of 100 microliters of 13C Octanoic Acid breath test
Ratings of palatability | 5 minutes (VAS scales for palatability once following the consumption of the test meal. This will be done for all 3 test meals provided to the participant, on the 3 separate days)
  Palatability ratings are assessed using a 100 mm Visual Analogue Scales (VAS, scale 0-100).
Ad-libitum meal consumption | 20 minutes (consumption of the meal weighed once post consumption. This will be done for all 3 test meals provided to the participant, on the 3 separate days)
  Consumption of the ad-libitum meal is measured (g). Participants are instructed to eat until they feel comfortable full and are given 20 min to consume the meal.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Methven, Principal Investigator — University of Reading
Locations (1):
- Sensory Science Centre, Department of Food and Nutritional Science, University of Reading, Reading, Berkshire, United Kingdom, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however it is possible that some of the individual (unliked / non identifiable) data will be useful in a meta analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Norton V, Lignou S, Methven L. Influence of Age and Individual Differences on Mouthfeel Perception of Whey Protein-Fortified Products: A Review. Foods. 2021 Feb 16;10(2):433. doi: 10.3390/foods10020433. PMID 33669435
- [Background] Norton V, Lignou S, Bull SP, Gosney MA, Methven L. An Investigation of the Influence of Age and Saliva Flow on the Oral Retention of Whey Protein and Its Potential Effect on the Perception and Acceptance of Whey Protein Beverages. Nutrients. 2020 Aug 19;12(9):2506. doi: 10.3390/nu12092506. PMID 32825104
- [Background] Clegg ME, Tarrado Ribes A, Reynolds R, Kliem K, Stergiadis S. A comparative assessment of the nutritional composition of dairy and plant-based dairy alternatives available for sale in the UK and the implications for consumers' dietary intakes. Food Res Int. 2021 Oct;148:110586. doi: 10.1016/j.foodres.2021.110586. Epub 2021 Jul 3. PMID 34507731
- [Background] Clegg ME, Williams EA. Optimizing nutrition in older people. Maturitas. 2018 Jun;112:34-38. doi: 10.1016/j.maturitas.2018.04.001. Epub 2018 Apr 4. PMID 29704915